CLINICAL TRIAL: NCT02997852
Title: Biobehavioral Effects of Therapy Dog Visitation in Elderly Intensive Care Unit Patients: A Pilot and Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Sandra M Branson, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-SN-15-0169
Record Dates: First submitted 2016-12-15; First posted 2016-12-20 (Estimated); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Psychosocial Stress
Keywords: human-animal interaction
MeSH Terms: conditions — Human-Animal Interaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Therapy dog visitation (Experimental): The TDV will consist of a 10-minute visit from the same Faithful Paws animal handler and her dog. Each therapy dog meets obedience, temperament, and health standards appropriate to therapy dog visitation in hospital settings. The dog will be leashed and under control of the animal handler and the TDV will be casual and not restrict the handler with conversing, which is standard practice in TDV. Visual and tactile contact with the dog will be promoted by the animal handler. Per hospital protocol, the patient will be assisted in washing his/her hands before and after the TDV and the dog will be placed on the bed or remain at the bedside in close proximity allowing petting. A clean sheet will be placed over the patient when the dog is placed on the bed. The research staff will collect data before and after each arm of the study.
  Interventions: Behavioral: Therapy dog visitation
- Control (No Intervention): Usual care in the intensive care unit.

INTERVENTIONS:
Behavioral: Therapy dog visitation — The TDV will consist of a 10-minute visit from the same Faithful Paws animal handler and her dog. Each therapy dog meets obedience, temperament, and health standards appropriate to therapy dog visitation in hospital settings. The dog will be leashed and under control of the animal handler and the TDV will be casual and not restrict the handler with conversing, which is standard practice in TDV. Visual and tactile contact with the dog will be promoted by the animal handler. Per hospital protocol, the patient will be assisted in washing his/her hands before and after the TDV and the dog will be placed on the bed or remain at the bedside in close proximity allowing petting. A clean sheet will be placed over the patient when the dog is placed on the bed. The research staff will collect data before and after each arm of the study.
  Arms: Therapy dog visitation

SUMMARY:
The purpose of this study is to assess the preliminary efficacy of a 10-minute therapy dog visitation (TDV) in reducing biobehavioral stress responses.

ELIGIBILITY:
Inclusion Criteria:

* ≥50 years old
* able to provide consent and understand English
* able to complete study instruments

Exclusion Criteria:

* currently taking hormone replacement or steroidal anti-inflammatory medications,
* in contact precautions at facility,
* diagnosed with Addison's or Cushing's disease
* fears or phobias to dogs, or allergies to dogs.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-07-25 (Actual); Primary Completion 2018-02-26 (Actual); Study Completion 2018-02-26 (Actual)

PRIMARY OUTCOMES:
Change in stress as assessed by the Stress-Visual Analog Scale | immediately before TDV, immediately after TDV
  Stress will be measured using the Stress-Visual Analog Scale which is a tool used in intensive care unit (ICU) settings that consists of a small, unmarked 100mm ruler with endpoints labeled "none" and "as bad as it could be". Participants indicate how stressed they feel on the ruler, which yields a single subjective stress score between 0 and 100. The Stress visual analogue scale (VAS) demonstrates acceptable validity between the VAS and the Hospital Anxiety and Depression (HADS) total score with correlations of r = 0.65.
Change in Anxiety as assessed by the Faces Anxiety Scale | immediately before TDV, immediately after TDV
  Anxiety will be measured using the FACES Anxiety Scale, a brief single-item, five-point self-report scale commonly used in the ICU consisting of 5 faces representing an increased level of anxiety, where the first item represents a "no anxiety" face (Elkman & Friesen; 1975). The FACES Anxiety Scale is a commonly used instrument in the ICU and proposed by the American Association of Critical-Care Nurses and demonstrates acceptable criterion validity between the FACES Anxiety Scale and State Anxiety Inventory total score in ventilated and non-ventilated ICU patients with correlations of r =.70; p<0005.
Change in Mood as assessed by the Positive and Negative Affect Schedule | immediately before TDV, immediately after TDV
  Measures for mood (positive/negative affect) will be measured using the Positive and Negative Affect Schedule (PANAS). The PANAS is an established 20-item instrument that uses a 5-point Likert scale and includes single words that express negative and positive moods. The instructions on the instrument would be revised to state, "indicate how you feel right now" rather than "indicate how you felt in the last week." Sample answers include "excited", "scared", "nervous", and "enthusiastic," etc. (Craword & Henry, 2004).
Change in biological stress response as assessed by salivary cortisol levels | immediately before TDV, immediately after TDV
  Saliva samples will be assayed using standardized enzyme immunoassay (EIA) kits (Salimetrics, State Park: PA). For cortisol, intra-assay coefficient of variation (CV) ranges between 4%-7% and inter-assay CV ranges between 3%-11%. Sensitivity of the EIA kit is .0007 μg/mL.
Change in biological inflammatory stress responses as assessed by salivary C-reactive protein (CRP) levels | immediately before TDV, immediately after TDV
  Saliva samples will be assayed using standardized enzyme immunoassay (EIA) kits (Salimetrics, State Park: PA). For CRP, intra-assay CV ranges between 1.9%-5.9% and inter-assay CV ranges between 3.7%-11.2%. Sensitivity of the EIA kit is 10 pg/mL.
Change in biological inflammatory stress responses as assessed by salivary interleukin-1beta (IL-1β) levels | immediately before TDV, immediately after TDV
  Saliva samples will be assayed using standardized enzyme immunoassay (EIA) kits (Salimetrics, State Park: PA). For IL-1β, intra-assay CV ranges between 2-3% and inter-assay CV is 4.5%. Sensitivity of the EIA kit is 0.6 pg/mL.

SECONDARY OUTCOMES:
Attachment level to pets as assessed by the Pet Attitude Scale (PAS) | immediately before TDV
  Attachment to pets will be measured using the Pet Attitude Scale (PAS) Questionnaire. The PAS is considered a reliable instrument in the elderly with a Cronbach's alpha of 0.73.
Human-Animal Interaction as assessed by the Human-Animal Interaction Scale (HAIS) | immediately after TDV
  The Human-Animal Interaction Scale (HAIS) is a newly developed questionnaire designed to measure behavioral interactions between animal and human which predict beneficial effects to humans (Fournier, Letson, Laitalia, & Krog, 2015). The HAIS is a 26 item Likert Scale with 5 Likert response statements ranging from "not at all" to "a great deal" and is completed by the participant after the TDV.
Human-Animal Interaction as assessed by the HAIS observer questionnaire | immediately after TDV
  The HAIS observer questionnaire is a 24 item instrument completed by the research staff who quantifies behaviors with a percent or range in respect to the behavior observed.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra M Branson, PhD, MSN, RN, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States